CLINICAL TRIAL: NCT01812135
Title: A Double-blind and Randomized, Phase II -02 Study With Inactivated EV71 Vaccines in Healthy Infants
Brief Title: Safety and Immunogenicity of EV71 Vaccine With or Without Aluminum Adjuvant in Infants
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Based on the previous study results, inactivated EV71 vaccine with aluminum adjuvant was elected to be used for the efficacy Phase III study.
Sponsor: Sinovac Biotech Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: EV71-1001-II-02
Record Dates: First submitted 2013-03-13; First posted 2013-03-15 (Estimated); Last update posted 2021-07-29 (Actual); Status verified 2013-03

CONDITIONS: Infection, Viral, Enterovirus
MeSH Terms: conditions — Infections; Enterovirus Infections | interventions — Adjuvants, Pharmaceutic

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1: 400U EV71 vaccine without adjuvant (Experimental): 60 infants received 2 doses of 400U EV71 vaccine without aluminium hydroxide adjuvant 28 days apart
  Interventions: Biological: 400 U EV71 vaccine with adjuvant
- Group 2: 400U EV71 vaccine without adjuvant (Experimental): 60 infants received 1 doses of 400U EV71 vaccine without aluminium hydroxide adjuvant
  Interventions: Biological: 400 U EV71 vaccine with adjuvant
- Group 3: 400U EV71 vaccine with adjuvant (Experimental): 60 infants received 1 doses of 400U EV71 vaccine with aluminium hydroxide adjuvant
  Interventions: Biological: 400 U EV71 vaccine with adjuvant

INTERVENTIONS:
Biological: 400 U EV71 vaccine with adjuvant — 400 U EV71 vaccine contain 0.4 mg AL/0.5 ml aluminum hydroxide adjuvant
  Other Names: EV71 vaccine

SUMMARY:
A randomized, double-blind, phase II-02 clinical trial is to evaluate the safety and immunogenicity of an inactivated EV71 vaccine with or without aluminum adjuvant

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males and females, aged from 6 to 11 months old Health is determined by medical history, physical examination, laboratory examination and clinical judgment of the investigator
2. Provided legal identification for the sake of recruitment.
3. Subjects and/or parent(s)/legal guardian(s) are able to understand and sign informed consents.
4. Birth weight more than 2500 grams

Exclusion Criteria:

1. History of Hand-foot-mouth Disease
2. Subject that has allergic history of vaccine, or allergic to any ingredient of vaccine
3. Serious adverse reactions to vaccines such as anaphylaxis, hives, respiratory difficulty, angioedema, or abdominal pain
4. Congenital malformations or developmental disorders, genetic defects, or severe malnutrition
5. Epilepsy, seizures or convulsions history, or family history of mental illness
6. Autoimmune disease or immunodeficiency, or parents, brothers and sisters have autoimmune diseases or immunodeficiency
7. History of asthma, angioedema, diabetes or malignancy
8. History of thyroidectomy or thyroid disease that required medication within the past 12 months
9. Bleeding disorder diagnosed by a doctor (e.g. factor deficiency, coagulopathy, or platelet disorder requiring special precautions) or significant bruising or bleeding difficulties with IM injections or blood draws
10. Asplenia, functional asplenia or any condition resulting in the absence or removal the spleen
11. Acute illness or acute exacerbation of chronic disease within the past 7 days
12. Any history of immunosuppressive medications or cytotoxic medications or inhaled corticosteroids within the past six months (with the exception of corticosteroid nasal spray for allergic rhinitis or topical corticosteroids for an acute uncomplicated dermatitis)
13. History of any blood products within 3 months
14. Administration of any live attenuated vaccine within 28 days
15. Administration of subunit or inactivated vaccines ,e.g., pneumococcal vaccine, or allergy treatment within 14 days
16. Axillary temperature > 37.0 centigrade before vaccination
17. Abnormal laboratory parameters before vaccination
18. Any medical, psychiatric, social condition, occupational reason or other responsibility that, in the judgment of the investigator, is a contraindication to protocol participation or impairs a volunteer's ability to give informed consent

Ages: 6 Months to 11 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2011-09; Primary Completion 2011-11 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Neutralization antibody geometric mean titer in infants 28 days after immunization with 400U vaccine with or without aluminium hydroxide adjuvant | 2 months
  Primary immunogenicity end point were geometric mean titer of neutralization antibody againt EV71 virus >= 1:8

SECONDARY OUTCOMES:
The rates and severity of solicited and unsolicited adverse events in infants following immunization as a Measure of Safety and Tolerability | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Yan-pin Li, MD, Principal Investigator — Guangxi Centers for Disease Control and Prevention
Locations (1):
- GuangXi Center for Diseases Control and Prevention, Nanning, Guangxi, China